CLINICAL TRIAL: NCT07103057
Title: ACCESS HCM: Real World Evidence for Artificial-Intelligence-assisted Screening and Access to Care for HCM - A Multi-Site Registry
Brief Title: VIZ ACCESS HCM - Multi-Site Registry
Status: Recruiting | Type: Observational
Sponsor: Viz.ai, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Viz-HCM-10
Record Dates: First submitted 2025-05-13; First posted 2025-08-05 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Artificial Intelligence; HCM
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (5):
- Cohort 1- Newly Diagnosed Patients: This cohort will consist of individuals who are newly diagnosed with HCM after the site began using Viz HCM. These patients will serve as a key population to assess the AI tool's impact on diagnoses, timeliness, and subsequent initiation of treatment. Data collected will include pre-diagnostic clinical indicators, diagnostic pathways, and treatment decisions following diagnosis. This cohort will begin to describe patient access to care and the clinical outcomes following a new HCM diagnosis in an AI-augmented clinical workflow.
  Interventions: Device: Viz HCM
- Cohort 2 - Previously Diagnosed Patients: Patients in this cohort will have an existing diagnosis of HCM prior to the start of using Viz HCM. This group will allow for the evaluation of how the AI tool may influence ongoing management strategies, such as treatment adjustments, monitoring practices, risk stratification, and clinical outcomes. The cohort will also help assess whether the AI tool facilitates optimization of care by identifying missed opportunities or previously unrecognized complications.
  Interventions: Device: Viz HCM
- Cohort 3 - Suspected and Not Diagnosed Patients: This cohort will include patients who were suspected by Viz HCM users of having underlying HCM, but clinical work-up sufficient to produce a diagnosis of HCM (including imaging and/or genetic testing) did not occur within the data collection period. Data collected will focus on diagnostic pathways, attempts made to coordinate care, and categorical barriers to care.
  Interventions: Device: Viz HCM
- Cohort 4 - Unlikely HCM: This cohort will look at a subset of randomly selected patients who are suspected by Viz HCM of having underlying HCM but are moved to the subgroup 'Unlikely HCM' within the Viz app/web by a clinician. After 1 year of study enrollment, a list will be created by Viz and shared with study teams for collection of additional minimal data including age, sex, reason for unlikely HCM (via chat), demographics (race, ethnicity) and reason for ECG.
  Interventions: Device: Viz HCM
- Cohort 5 - Alerts Not Reviewed: This cohort will look at a subset of randomly selected patients who are suspected by Viz HCM of having underlying HCM, but the alert is never reviewed by a clinician. After 1 year of study enrollment, a list will be created by Viz and shared with study teams for collection of additional minimal data including age, sex, demographics (race, ethnicity) and reason for ECG.
  Interventions: Device: Viz HCM

INTERVENTIONS:
Device: Viz HCM — Viz HCM is a Software as a Medical Device (SaMD) intended to receive 12-lead ECG recordings collected as part of a routine clinical assessment and analyze them in parallel to the standard of care. The device uses a machine learning based algorithm to analyze 12-lead ECGs and identify ECGs with suspected HCM.

SUMMARY:
To describe the clinical, economic, and population characteristics of newly diagnosed, previously diagnosed, and suspected patients evaluated by Viz HCM. HCM is underdiagnosed in the community and AI algorithms have been developed as screening tools. However, it is not well understood how to best integrate AI screening tools and their potential impact.

ELIGIBILITY:
All Cohorts

* Patients aged 18+ years at time of arrival to healthcare facility
* Patients with a resting 12-lead digital electrocardiogram (ECG) that is flagged by Viz HCM for HCM suspicion

Additional cohort-specific criteria:

Cohort 1 - Newly Diagnosed Patients

* Patients have been diagnosed with HCM after the Viz HCM implementation
* Written informed consent is obtained prior to data collection

Cohort 2 - Previously Diagnosed Patients ● Prior diagnosis of HCM as evidenced by clinical diagnosis documentation prior to Viz HCM implementation

Cohort 3 - Suspected and Not Diagnosed Patients

● Patients did not receive sufficient clinical workup for HCM diagnosis confirmation

Cohort 4 - Unlikely HCM ● Patient ECG moved to 'Unlikely HCM' group within Viz by site study staff following HCM alert review

Cohort 5 - Alerts Not Reviewed

● HCM alert not reviewed by site study staff during study enrollment period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who have an ECG that has been flagged by Viz HCM.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Clinical characteristics of Viz HCM AI screening on HCM diagnosis | Up to 3 years
  To describe the clinical characteristics of patients who were alerted for suspected HCM by an AI-based ECG tool and newly diagnosed, previously diagnosed, or suspected for HCM.
Clinical characteristics of Viz HCM AI screening on medical workup. | Up to 3 years
  To describe the clinical characteristics of medical workup for patients who were alerted for suspected HCM by an AI-based ECG tool and newly diagnosed, previously diagnosed, or suspected for HCM.
Clinical characteristics of Viz HCM AI screening on treatment plans. | Up to 3 years
  To describe the clinical characteristics of treatment plans for patients who were alerted for suspected HCM by an AI-based ECG tool and newly diagnosed, previously diagnosed, or suspected for HCM.
Clinical characteristics of Viz HCM AI screening on closed care pathways | Up to 3 years
  To describe the clinical characteristics of closed care pathways (patients diagnosed who receive treatment) for patients who were alerted for suspected HCM by an AI-based ECG tool and newly diagnosed, previously diagnosed, or suspected for HCM.
Population evaluation for access to care by socioeconomic status at the time of diagnosis. | Up to 3 years
  To describe HCM access to care by socioeconomic status at the time of diagnosis.
Population evaluation for access to care by clinical stage of HCM at time of diagnosis. | Up to 3 years
  Population evaluation for access to care by clinical stage of HCM at time of diagnosis.
Healthcare utilization and health economic outcomes- medical clinic visits | Up to 3 years
  To describe healthcare utilization and economic outcomes as captured by medical clinic visits, associated testing (e.g., echocardiogram, cardiac MRI, laboratory and genetic screening), hospitalization, and ICD placement for primary and secondary prevention for sudden cardiac death.
Health economics outcome as captured by associated testing modalities | Up to 3 years
  To describe healthcare utilization and economic outcomes as captured by associated testing
Health economics outcome as captured by hospitalization data | Up to 3 years
  To describe healthcare utilization and economic outcomes as captured by hospitalization data
Health economics outcome as captured by ICD placement data | Up to 3 years
  To describe healthcare utilization and economic outcomes as captured by ICD placement for primary and secondary prevention for sudden cardiac death.

SECONDARY OUTCOMES:
Implementation science - percentage of alerts viewed | Up to 2 years
Implementation science - number of active users over time | Up to 2 years
Implementation science - reasons for user-indicated actions, where documented | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Milind Desai, MD, Principal Investigator — The Cleveland Clinic
Locations (3):
- United States (3):
  - Emory University, Atlanta, Georgia
  - North Shore University Health System, Evanston, Illinois
  - Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No